CLINICAL TRIAL: NCT06971224
Title: NADream: Effects of Nicotinamide Adenine Dinucleotide Supplementation on Sleep Quality in Healthy Individuals: A Randomized Controlled Pilot Study
Brief Title: NADream: Effects of Nicotinamide Adenine Dinucleotide Supplementation on Sleep Quality in Healthy Individuals
Acronym: NADream
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/849242
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Sleep
Keywords: Sleep; Nicotinamide Riboside; NR; Nicotinamide adenine dinucleotide; NAD; Polysomonography; PSG
MeSH Terms: interventions — nicotinamide-beta-riboside; NAD

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo-controlled study with a duration of 8 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and all care providers and investigators are blinded during the trial and during data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside (NR) (Experimental): Nicotinamide Riboside (NR) administered in doses of 1000 mg twice daily for the duration of the trial (8 weeks).
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- Placebo (Other): Placebo, no active ingredients. Administered in tablet form twice daily for the duration of the trial (8 weeks).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — 2000 mg NR daily.
  Other Names: Nicotinamide adenine dinucleotide (NAD)
  Arms: Nicotinamide Riboside (NR)
Other: Placebo — Placebo tablet identical in taste, shape and appearance to NR tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evalue the effects of nicotinamide adenine dinucleotide (NAD) supplementation (nicotinamide riboside (NR) form) on sleep in healthy adults compared to a placebo. NAD is important for brain health and energy balance and a proposed explanation for its effect on sleep is that NAD supplementation restores the neurophysiological capacity of the brain to 'rest' during sleep. If this is the case, we expect the administration to result in improvements in sleep quality (and most likely sleep quantity) compared to placebo. Participants will receive either NAD supplementation or a placebo and their sleep will be measured to detect any differences between the two groups.

DETAILED DESCRIPTION:
Nicotinamide adenine dinucleotide (NAD+) is important for regulating cellular energy metabolism, mitochondrial function, and circadian rhythms, which are key processes involved in the sleep-wake cycle and sleep regulation. Nicotinamide riboside (NR) supplementation has been shown to elevate NAD+ levels in humans. Higher NAD+ levels may support better sleep by restoration of mitochondrial efficiency and reducing oxidative stress.

As people age, there is evidence of a decline in NAD+ levels, which may lead to mitochondrial dysfunction, oxidative stress, and disruptions in circadian rhythms. These changes can negatively affect sleep architecture and reduce sleep quality. Impaired NAD+ metabolism has been linked to problems with the molecular clock, which regulates circadian timing through effects on sirtuin activity and clock genes such as BMAL1. NAD+ also supports brain metabolism by maintaining mitochondrial function, promoting neuroprotection, regulating redox balance, and reducing neuroinflammation. By restoring NAD+ levels, NR supplementation may help improve mitochondrial efficiency, decrease oxidative damage, and enhance sleep-related cellular maintenance. NR may also support synchronization of circadian rhythms, further promoting healthy sleep. Its effects also include modulating neuroinflammatory pathways and strengthening cellular resilience against oxidative stress, both of which are essential for maintaining cognitive functions and neural plasticity during sleep.

The NADream study will test whether NR supplementation can improve both objective and subjective measures of sleep in healthy adults. Sleep will be assessed using polysomnography (PSG), the gold standard for objective sleep measurement, along with actigraphy, Somnofy sleep monitoring, and the Pittsburgh Sleep Quality Index (PSQI). This study will be a randomized, placebo-controlled, double-blind, parallel-group design. Participants will be randomly assigned to receive ether NR or a placebo for 8 weeks. The findings from this study will help determine whether NR supplementation could be a viable therapeutic option to explore further in this area.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 40 to 60 years of age inclusive, at the time of signing the informed consent.
* Male or female.
* Participants who are healthy as determined by medical evaluation including medical history and physical examination.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the study protocol.
* Self-reported normal sleep patterns, assessed by Pittsburgh sleep quality index (PSQI; cutoff ≤ 5).
* No current use of sleep medications or supplements.
* Able to wear polysomnographic equipment and actigraphy during nighttime.

Exclusion Criteria:

* History of sleep disorders (e.g. insomnia, sleep apnea).
* Abnormal findings on PSG, such as sleep related breathing disorders (apnea-hypopnea index (AHI) ≥ 5), sleep related movement disorders (periodic limb movement index (PLMI) ≥ 15, and parasomnias (like REM sleep behavior disorder (RBD)).
* Chronic use of alcohol, tobacco, or medications affecting sleep.
* Significant psychiatric or medical conditions (including neurological, heart, lung, or sleep disorders/diseases).
* Travelled >1 time zone and night work <1 month before study, or during the study.
* Extreme chronotype according to the Composite Morningness Questionnaire (evening type; <22 and morning type >44).
* Pregnancy.
* Breastfeeding.
* Supplements resulting in > 20 mg daily of nicotinamide riboside, nicotinamide mononucleotide (NMN), niacin (vitamin B3, nicotinic acid amide or other vitamin B3 analogues) less than 3 months prior to randomization.
* Participation in other clinical trials last 3 months.
* Deemed ineligible by lead principal investigator.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of NAD supplementation on objective sleep parameters via polysomnography (PSG). | From enrollment to the end of treatment at 8 weeks.
  The primary endpoint is the change in electrophysiological slow-wave activity (SWA; 0.5 - 4.0 Hz) per 60 minutes, measured by EEG, from baseline to week 8 between the 2000 mg NR and placebo groups.

SECONDARY OUTCOMES:
The secondary endpoints are to evaluate the effect of NAD supplementation on objective sleep parameters via polysomnography (PSG). | From enrollment to the end of treatment at 8 weeks.
  Slow wave energy (SWE) during sleep. Accumulated SWA as a putative homeostatic marker of sleep drive.
EEG power | From enrollment to the end of treatment at 8 weeks.
  EEG power for each sleep stage in 1 Hz bins from 1 to 20 Hz.
Arousals during sleep. | From enrollment to the end of treatment at 8 weeks.
  Arousals during sleep (abrupt cortical awakenings lasting >3 seconds).
Theta activity. | From enrollment to the end of treatment at 8 weeks.
  Theta activity (5 - 8 Hz) during REM sleep, as a marker of REM sleep quality.
Time in bed (TIB). | From enrollment to the end of treatment at 8 weeks.
  Time in bed (TIB, in minutes). Total time the person is laying down in bed.
Sleep onset latency (SOL). | From enrollment to the end of treatment at 8 weeks.
  Sleep onset latency (SOL, in minutes). Length of time from full wakefulness to sleep.
Total sleep time (TST). | From enrollment to the end of treatment at 8 weeks.
  Total sleep time (TST, in minutes). Total time the person sleeps.
Sleep architecture. | From enrollment to the end of treatment at 8 weeks.
  Sleep architecture: time spent in non-rapid eye movement (NREM) stages and REM sleep, particularly the more restorative and deep sleep (stage N3/slow wave sleep) will be examined.
Wake after sleep onset (WASO). | From enrollment to the end of treatment at 8 weeks.
  Wake after sleep onset (WASO, in minutes). Periods of wakefulness after defined sleep onset.
Sleep efficiency (SE). | From enrollment to the end of treatment at 8 weeks.
  Sleep efficiency (SE) (time asleep/TIBx100)

OTHER OUTCOMES:
Cognitive function. | From enrollment to the end of treatment at 8 weeks.
  Specific subtests of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Blood biomarkers. | From enrollment to the end of treatment at 8 weeks.
  Blood samples for oxidative stress biomarkers, including inflammatory profiles (CRP, IL-6, TNF-alpha).
NAD metabolome. | From enrollment to the end of treatment at 8 weeks.
  NAD metabolome in blood, measured by LC-MS metabolomics and/or NADMED assay.
Blood samples. | From enrollment to the end of treatment at 8 weeks.
  Blood samples for biobank.
Subjective sleep parameters using validated questionnaires. | From enrollment to the end of treatment at 8 weeks.
  Pittsburg Sleep Quality Index (PSQI), Chalder fatigue questionnaire (CFQ), Karolinska Sleepiness Scale (KSS), Composite Morningness Questionnaire (CMQ).
Objective activity patterns tracked by non-invasive device. | From enrollment to the end of treatment at 8 weeks.
  Activity/inactivity pattern across successive days derived by actigraphy (Axivity).
Objective sleep patterns tracked by non-invasive device. | From enrollment to the end of treatment at 8 weeks.
  Sleep monitoring successive days derived by Somnofy (Vital Things AS).

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, PhD, Study Director — Haukeland University Hospital; Katarina Lundervold, MD, Principal Investigator — University of Bergen; Janne Grønli, PhD, Principal Investigator — University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No